CLINICAL TRIAL: NCT02376270
Title: The Effects of Pectin on Aging-related Changes in Intestinal Barrier Function, Immune Function and Microbial Composition
Brief Title: Pectin, Aging and Intestinal Barrier Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 143055
Record Dates: First submitted 2015-02-19; First posted 2015-03-03 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2015-10

CONDITIONS: Healthy Young Adults; Healthy Elderly
MeSH Terms: interventions — Pectins; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Pectin (Experimental): This group will receive 7.5 grams of pectin supplements twice daily for four weeks.
  Interventions: Dietary Supplement: Pectin
- Maltodextrin (Placebo Comparator): This group group will receive 7.5 grams of maltodextrin supplements twice daily for four weeks.
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Pectin — This group will receive 7.5 grams of pectin supplements twice daily for four weeks.
  Arms: Pectin
Dietary Supplement: Maltodextrin — This group will receive 7.5 grams of maltodextrin supplements twice daily for four weeks.
  Arms: Maltodextrin

SUMMARY:
The population is aging worldwide, which requires more attention to health needs and leads to a dramatic increase in health care costs. Prevention or delay of onset of disorders associated with aging is needed. Dietary intake of pectin, a dietary fiber, may have beneficial effects on gut health parameters, i.e. intestinal barrier function, immune function and microbial composition. As intestinal barrier function may be compromised in the elderly we will investigate whether the effects of pectin on selected parameters of gut health differ between young vs. older individuals. The primary objective of this study is to investigate the effects of aging on pectin-induced changes in intestinal permeability. Furthermore, this study has seven secondary objectives. This study conforms to a randomized, double-blind and placebo-controlled design including two parallel arms.The study population consists of Healthy human volunteers (male and female), 18-40 and 65-75 years old, BMI 20-30 kg/m2. One group will receive 7.5 grams of pectin supplements twice daily for four weeks. A second group will receive 7.5 grams of placebo supplements twice daily for four weeks. Before and after the supplementation period, several measurements will take place. The main study parameter is the change in urinary sugar excretion ratio before and after the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Based on medical history and previous self-admitted examination, no gastrointestinal complaints can be defined.
* Age between 18 - 40 years and 65 - 75 years.
* Body Mass Index (BMI) between 20 and 30 kg/m2. Normal BMI has been chosen because obesity is associated with an altered microbial composition and increased intestinal permeability.

Exclusion Criteria:

* History of severe cardiovascular, respiratory, urogenital, gastrointestinal/ hepatic, hematological/immunologic, HEENT (head, ears, eyes, nose, throat), dermatological/connective tissue, musculoskeletal, metabolic/nutritional, endocrine, neurological diseases, allergy, major surgery and/or laboratory assessments which might limit participation in or completion of the study protocol.
* Use of proton-pump inhibitors, nonsteroidal anti-inflammatory drugs and/or vitamin supplementation, within 14 days prior to testing. Use of other medication will be reviewed by a medical doctor, who will decide on in- or exclusion based on the drug(s) used.
* Administration of probiotic or prebiotic supplements, investigational drugs or participation in any scientific intervention study which may interfere with this study (to be decided by the principle investigator), in the 90 days prior to the study
* Use of antibiotics in the 90 days prior to the study.
* Abdominal surgery interfering with gastrointestinal function, upon judgment of the principle investigator).
* Pregnancy, lactation.
* Excessive alcohol consumption (>20 alcoholic consumptions per week).
* Smoking.
* Blood donation within 3 months before or after the study period.
* Self-admitted human immunodeficiency virus-positive state.
* History of side effects towards intake of prebiotic supplements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Sugar recovery in urine, as indicator of intestinal permeability | Change from Baseline to after 4 weeks of intervention

SECONDARY OUTCOMES:
Tight junction structure and proteins in colonic biopsies, as indicator of intestinal barrier function | After 4 weeks of intervention
Ussing chamber experiments in colonic biopsies, as indicator of intestinal barrier function | After 4 weeks of intervention
Histology in colonic biopsies, as indicator of intestinal barrier function | After 4 weeks of intervention
MiR-29a in colonic biopsies, as indicator of intestinal barrier function | After 4 weeks of intervention
Zonulin in blood plasma, as indicator of intestinal barrier function | Change from Baseline to after 4 weeks of intervention
Immune infiltration cells in colonic biopsies, as indicator of immune system performance | After 4 weeks of intervention
T-cells and Natural Killer cells in blood plasma, as indicator of immune system performance | Change from Baseline to after 4 weeks of intervention
Cytokines Interleukin-10 and Interleukin-12 in blood plasma, as indicator of immune system performance | Change from Baseline to after 4 weeks of intervention
C-reactive protein in blood serum, as indicator of immune system performance | Change from Baseline to after 4 weeks of intervention
Secretory Immunoglobulin A in blood serum, as indicator of immune system performance | Change from Baseline to after 4 weeks of intervention
Microbial composition in luminal content and feces | Change from Baseline to after 4 weeks of intervention
Short-chain fatty acids in luminal content and feces, as indicator of microbial function | Change from Baseline to after 4 weeks of intervention
Volatile organic compounds in exhaled air, as indicator for metabolite production | Change from Baseline to after 4 weeks of intervention
Symptom diary questionnaire, as indicator of digestive parameters | Change from three days prior to the supplementation period to three days during the last week of the supplementation period
Stool frequency and consistency questionnaire, as indicator of digestive parameters | Change from Baseline to after 4 weeks of intervention
Gastrointestinal Symptom Rating Scale questionnaire, as indicator of digestive parameters | Change from Baseline to after 4 weeks of intervention

CONTACTS AND LOCATIONS:
Overall Officials: A.A.M. Masclee, Professor, Principal Investigator — Department of Internal Medicine, Division of Gastroenterology-Hepatology
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands